CLINICAL TRIAL: NCT05612412
Title: Bone Metabolic Responses to Morning Versus Evening Exercise
Brief Title: Exercise for Better Bones - Day or Night?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GFHNRC154
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Exercise (Experimental): Morning exercise session
  Interventions: Other: Morning Exercise
- Evening Exercise (Experimental): Evening exercise session
  Interventions: Other: Evening Exercise

INTERVENTIONS:
Other: Morning Exercise — Standardized treadmill exercise session starting at approximately 0700
  Arms: Morning Exercise
Other: Evening Exercise — Standardized treadmill exercise session starting at approximately 1800
  Arms: Evening Exercise

SUMMARY:
The purpose of this study is to find out if moderate exercise at different time during the day (early morning vs early evening) affects biomarker CTX of bone health in normal to overweight postmenopausal women.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate whether the daily timing of exercise affects bone turnover markers in postmenopausal women. Results from this clinical trial will provide valuable information to support guidelines of physical activity for people to improve musculoskeletal health, especially post-menopausal women. The scientific questions that will be investigated are:

1. What are the acute effects of the daily timing of exercise on serum concentrations of bone turnover markers and 24-h total urinary calcium excretion?
2. Are differences in initial exercise-induced responses of bone turnover markers and urinary Ca excretion maintained across two weeks of exercise training?

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women within 1-10 yr after menopause
* BMI 18.5-29.9 kg/m2
* Healthy as determined by a screening physical examination and blood chemistry related to thyroid, liver, kidney, and lipid profile within normal range
* No osteoporosis as determined by dual energy x-ray absorptiometry (DEXA) scan at femoral neck or total spinal region
* No regular exercise for more than 30 minutes a day on more than 2 days a week and no physically active employment, such as maintenance and repair or delivery worker
* No regular use of medications known to interfere with calcium and bone metabolism from 6 weeks prior to the study to the end of study such as medications for heartburn, reflux, H2 blockers, diuretics, etc. such as antacids, Maalox, Pepcid AC, Nexium, Diuril, etc.
* Weight stable (within 5 lbs change) for at least 3 months prior to the start of the study
* Willing to maintain usual lifestyle and activities including the same wake-sleep schedule (go to sleep between 10:00 p.m. and midnight with an average 6-8 hours of sleep time)
* Refrain from the use of alcohol and nicotine (for example, cigarettes, cigars, and e-cigarettes) for the length of the study
* Able and willing to perform moderate intensity exercise without contraindications as determined by the Physical Activity Readiness Questionnaire
* Willing and able to stop any nutritional supplements including vitamin D supplements and calcium-containing medications (for instance, calcium-carbonate antacids)
* Willing not to use tanning booths during the study or not to travel to locations with a tropical climate two weeks prior to the study or during the washout period

Exclusion Criteria:

* Hypertension with resting blood pressure higher than systolic 140 and diastolic 90 mmHg
* Within past 6 weeks, had nutrition supplements or medications known to affect calcium metabolism and appetite such as Antacids, Megace, antacids, heartburn, reflux, H2 blockers, diuretics, etc.
* Allergy to any food ingredients used in the provided diet
* Any disorders affecting nutrient absorption or metabolism, such as cystic fibrosis, lactose intolerance, celiac disease, etc.
* Any sleep disorders such as sleep apnea or regular use of an over-the-counter melatonin supplement
* Diabetes or taking medications known to affect bone such as Actos, Avandia, Invokana, etc.
* Engaged in moderate to vigorous exercise or regular exercise for more than 30 minutes/day on more than 2 days/week within past 6 weeks
* Repeated non-compliance with completing prescribed exercise sessions
* Within past 6 weeks, used tanning booths or traveled to location with a tropic climate
* Use of antibiotics (Amoxicillin, doxycycline, etc.), nonsteroidal anti-inflammatory drugs (aspirin, Celebrex, etc.), or probiotics (Lactobacillus, Bifidobacterium) within the past 6 weeks
* Irritable bowel syndrome, inflammatory bowel disease, or not having a bowel movement three days or longer

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in serum C-terminal telopeptide of type 1 collagen (CTX) | Day 1, Day 15
  Test the differences in morning peak serum CTX following one bout of exercise per day for 10 days over a two-week period in either the early morning or the evening.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Cao, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT05612412/ICF_000.pdf